CLINICAL TRIAL: NCT00863421
Title: Prevalence, Incidence and Clinical Characteristics of Sleep Disordered Breathing in Patients With Stable Chronic Heart Failure
Brief Title: Sleep Disordered Breathing in Patients With Chronic Heart Failure
Acronym: VISIFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology (Network)
Responsible Party: Arschang Valipour, M.D., FCCP, Ass. Prof, Ludwig Boltzmann Institute for COPD Research
Other Study IDs: VISIFA 08-058-0508
Record Dates: First submitted 2009-03-15; First posted 2009-03-18 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Sleep-disordered Breathing; Chronic Heart Failure
Keywords: Sleep disordered breathing; Prevalence; Chronic heart failure; Incidence; Sleep apnea; Cheyne-Stokes-Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Only few prospective studies systematically investigated the prevalence of sleep disordered breathing in patients with stable chronic heart failure. Furthermore there is no report on the incidence rate of sleep disordered breathing in this population. This is a prospective multi-centre study of sleep-disordered breathing in 200 patients with stable moderate-to-severe chronic heart failure. Eligible patients will undergo overnight full-night polysomnography, lung function testing, laboratory measurements, and hemodynamic recordings. Measurements will be repeated at 6 months interval for a follow-up period of two years irrespective of the presence or absence of sleep disordered breathing. The primary outcome variable for this study is the prevalence of sleep disordered breathing in the study population. Secondary outcome variables include the 2-year incidence rate of sleep disordered breathing, quality of life measurements, exercise capacity, sleep quality, hemodynamic measurements, and laboratory markers of neurohumoral activation, systemic inflammation, and endothelial function in the study population.

DETAILED DESCRIPTION:
Chronic heart failure is a complex clinical syndrome that can result from any structural or functional cardiac or non-cardiac disorder that impairs the ability of the heart to respond to physiological demands for increased cardiac output. Chronic heart failure is characterised by symptoms such as exertional breathlessness and fatigue, and signs of fluid retention as well as signs associated with the underlying cardiac disorder. Patients with chronic heart failure suffer from reduced quality of life and a significantly higher risk of morbidity and mortality.

There is cumulating evidence of a high prevalence of sleep breathing disorders in both patients with acute and chronic heart failure. Most of these reports, however, suffer from important limitations including small sample size, retrospective study design, and/or use of pulse-oximetry or cardio-respiratory polygraphy to screen for sleep disordered breathing rather than full-night polysomnography. Hence, previous studies may have underestimated the full scale of concomitant sleep disordered breathing in patients with chronic heart failure. Furthermore, to the best of our knowledge, there is no report on the incidence of sleep disordered breathing in patients with chronic heart failure.

In this context the presence of sleep disordered breathing in patients with chronic heart failure has important prognostic relevance. Pathophysiological effects of sleep apnea include intermittent hypoxia, sympathetic hyperactivity, systemic inflammation, and sleep fragmentation. These factors may contribute to the worsening of cardiac function and explain the reportedly higher risk of cardiac morbidity and mortality in patients with both chronic heart failure and concomitant sleep disordered breathing. Accordingly, the aims of the present study are three-fold. First, to investigate the prevalence of sleep breathing disorders in patients with stable moderate-to-severe chronic heart failure using the diagnostic gold standard of full-night-polysomnography. Second, to assess the two-year incidence of sleep disordered breathing in patients with chronic heart failure. Third, to identify potential risk factors associated with the presence or absence of sleep disordered breathing in patients with chronic heart failure. The latter will be assessed by using lung function measurements, hemodynamic parameters, and laboratory markers of neurohumoral activation, systemic inflammation, and endothelial function in patients with chronic heart failure.

For this purpose 200 patients with stable moderate-to-severe chronic heart failure will be studied during a 2 year-period. Patients with chronic heart failure will be screened for eligibility during their regular visits at 4 independent heart failure outpatients clinic in Vienna. Eligible patients will undergo full-night-polysomnography, lung function testing, non-invasive hemodynamic monitoring, a six minute-walking-test, and laboratory measurements at 6 months intervals for a total of 2 years (4 visits).

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic heart failure(NYHA II-IV), defined as

  * a condition diagnosed for at least 6 months prior to inclusion under maximally tolerated medical therapy
  * without any relevant changes to symptoms or medication during the 8 weeks prior to inclusion
  * by the absence of any hospitalizations during the previous 3 month
* Ejection fraction equal or below 35%
* Age between 18 and 80 years

Exclusion Criteria:

* Instable angina pectoris
* Acute coronary syndrome within the last 6 months
* Cerebrovascular events (TIA, PRIND, stroke) within the last 12 months
* Primary pulmonary hypertension(systolic PAP > 45 mmHg)
* Congenital heart failure
* Primary heart valve disease
* Regular use of benzodiazepines, other sedatives, or opiate derivatives
* Severe renal(s-creatinine > 3 mg/dl) and/or liver disease(GPT > 3xULN)
* Clinically relevant affections of the central nervous system(e.g.epilepsy, multiple sclerosis,...)
* Known moderate to severe chronic obstructive pulmonary disease(FEV1/(F)VC < 70% und FEV1 < 50% Soll) or restrictive lung disease with total lung capacity < 70%
* Untreated hormonal disease(e.g.hypothyreosis,....)
* Daily alcohol consumption with more than 60g alcohol per day for men and more than 30g alcohol per day for women
* Implantation of a pacemaker or ICD within the previous 6 months
* St.p. aortocoronary bypass surgery or lung resection within the previous 12 month
* Women of child-bearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from 4 independent heart failure outpatient clinics in Vienna.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disordered breathing in patients with stable chronic heart failure | 2 years

SECONDARY OUTCOMES:
2-year-incidence of sleep disordered breathing in patients with stable chronic heart failure | 2 years
Prevalence of lung function abnormalities in patients with stable chronic heart failure | 2 years
Quality of Life in patients with and those without sleep disordered breathing using the Minnesota Living With Heart Failure Questionnaire and the SF-36. | 2 years
Sleep Quality in patients with and those without sleep disordered breathing using the Pittsburgh Sleep Quality Index, the Sleep Disorders Questionnaire, and the Functional Outcome of Sleep Questionnaire | 2 years
Exercise capacity in meters in the total study population using the 6-Minute-Walking-Test distance | 2 years
Pro brain natriuretic peptide, C-reactive protein, tumor-necrosis-factor alpha, interleukin-6, asymmetric dimethylarginine, vascular endothelial growth factor | 2 years
Measurements of cardiac output, heart rate variability, and baroreceptor sensitivity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, M.D., Principal Investigator — Ludwig Boltzmann Institute for COPD
Locations (1):
- Otto Wagner Hospital, Vienna, Vienna, Austria